CLINICAL TRIAL: NCT04511221
Title: BacterioPHAGE for Gastrointestinal Health 2 Study
Acronym: PHAGE2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Responsible Party: Principal Investigator, Tiffany Weir, Associate Professor of Food Science and Human Nutrition, Colorado State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 19-9145H
Record Dates: First submitted 2020-08-07; First posted 2020-08-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Mild Gastrointestinal Symptoms in Healthy Adults
Keywords: gastrointestinal; probiotic; bacteriophage; Bifidobacterium animalis subspecies lactis

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded, placebo controlled, parallel arm
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Treatment capsules are provided by Deerland Enzymes in coded packaging. Participants, investigators, and data assessors will not be provided the key to the codes. Once all data is entered and analyzed, the keys will be provided by Deerland.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): 15 mg capsule containing rice maltodextrin and medium chain coconut triglycerides
  Interventions: Other: Placebo
- Bifidobacterium animals subsp. lactis BL04 (Active Comparator): 15 mg capsule containing 1x 10^9 CFU Bifidobacterium animals subsp. lactis BL04 with rice maltodextrin and medium chain coconut triglycerides as a filler material
  Interventions: Dietary Supplement: Bifidobacterium animals subsp. lactis BL04
- Bifidobacterium animals subsp. lactis BL04+PreforPro (Experimental): 15 mg capsule containing 1x 10^9 CFU Bifidobacterium animals subsp. lactis BL04 and 1x10^6 PFU of PreforPro (Commercial phage preparation) with rice maltodextrin and medium chain coconut triglycerides as a filler material
  Interventions: Dietary Supplement: Bifidobacterium animals subsp. lactis BL04+PreforPro

INTERVENTIONS:
Dietary Supplement: Bifidobacterium animals subsp. lactis BL04+PreforPro — One 15mg capsule taken orally each day
  Arms: Bifidobacterium animals subsp. lactis BL04+PreforPro
Dietary Supplement: Bifidobacterium animals subsp. lactis BL04 — One 15mg capsule taken orally each day
  Arms: Bifidobacterium animals subsp. lactis BL04
Other: Placebo — One 15mg capsule taken orally each day
  Arms: Placebo

SUMMARY:
The BacterioPHAGE for Gastrointestinal Health-2 study is designed to determine if a commercial bacteriophage product can increase the survival and efficacy of probiotic bacteria that will be concurrently administered. Bacteriophages may act as prebiotics, which are traditionally defined as indigestible dietary components that selectively enhance specific bacterial species in the intestines to confer a health benefit. In this study, the "prebiotic" is a unique combination of bacteriophages, or viruses that infect bacteria. These phages are generally regarded as safe for human consumption and are presumed to function by infecting pro-inflammatory E. coli strains in the gut. The removal of these strains alters the gut environment to allow growth of more favorable bacteria, and the lysis products of these E. coli may be assimilated by beneficial species to enhance their populations.The phage product, PreforPro, has shown to be effective in culture-based and animal studies, but its efficacy in increasing specific probiotic species has not been demonstrated in humans. The investigators have previously shown that PreforPro is both safe and tolerable in a human population and does not broadly disrupt the gut microbiota as would be seen with antibiotic treatment.

DETAILED DESCRIPTION:
The commercial bacteriophage preparation,PreforPro, is often found as an ingredient in commercial probiotcs, so the goal of the current study is to determine if PreforPro consumption concurrent with probiotic usage improves probiotic survival and activity. A secondary goal of this study is to assess various physiologic parameters to determine whether consumption of PreforPro with a probiotic offers any health benefits beyond those of consuming a probiotic alone. The investigators will examine whether consumption of the PreforPro product increases detectable numbers of co-consumed probiotics and improves parameters in clinical outcomes related to glucose and lipid metabolism, cardiovascular function, inflammation of the intestines, or physical symptoms of gastrointestinal distress.

To accomplish these research goals, the investigators will be seeking 200 male and female volunteers between 18-65 years old with BMI scores of 22 to 34.9. Recruitment will be by referral from local practitioners, email recruitment, and through word-of-mouth. Eligibility will be determined at the Colorado State University Food and Nutrition Clinical Research lab by a screening questionnaire and interview/assessment by the clinical coordinator. After securing consent, eligibility will be confirmed by taking anthropometric measures and participants falling within the BMI range will randomly be assigned to 1 of 3 treatment groups: (1) PreforPro+Bifidobacterium probiotic, (2) Bifidobacterium probiotic alone, or (3) placebo. Participants will consume the provided capsules daily for a period of four (4) weeks. Participants will be asked to visit the clinic at Visit 1 (Day 0) to pick up their supply of capsules and undergo sample collections (blood and stool) and analysis procedures, including weight/height, blood pressure, endothelial function analysis, gastrointestinal symptom screening, and blood and stool sample collection. At the end of the 4 week treatment period, all analyses will be repeated. This means that participants will undergo screening (either in person or by phone) and make a total of two (2) clinic visits during the study (baseline, and final visit). Participants will additionally be asked to complete two 24 hour dietary recalls prior to each clinic visit and track bowel movements using the Bristol Stool Scale throughout the study treatment period. All blood samples will be collected at Colorado State University by trained personnel. Fecal sample collection will be performed by the study participant with collection materials provided.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* 18-65 years old
* BMI 20 to 34.9

Exclusion Criteria:

* individuals less than 18 years of age or greater than 65 years of age
* outside of the BMI range of 20-34.9
* antibiotic or probiotic/prebiotic supplements within two months of the start of treatment
* use of statins, metformin, NSAIDs, MAO inhibitors, and botanical supplements that target the GI tract or gut microbiota
* current diagnosis of cancer, liver or kidney disease, gastrointestinal diseases, and metabolic disorders
* pregnant and breastfeeding women
* unable to adhere to the study requirements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal Symptoms | Four weeks
  A functional gastrointestinal questionnaire was used to assess pain and symptoms related to GI function, GI inflammation, Colon and small intestine pain
Bowel Function | Four weeks
  A record of all stools (using Bristol Stool Scale) was collected throughout the study
Microbiota Analysis | Four weeks
  16s sequencing and phage plating was conducted to assess phage activity and microbiota associated changes.

SECONDARY OUTCOMES:
Blood pressure | Four weeks
  Blood pressure will be measured on non-dominant arm using a Sphygmacor. Three consecutive measures will be taken after particioants have spent 5 minutes in a supine position.
Endothelial Function | Four Weeks
  Endothelial function will be measured using EndoPat technology and expressed as Reactive Hyperemia Index (RHI)
Plasma Lipids | Four weeks
  A single venous blood sample will be collected and 200 ul added to a Piccolo test
  cartridge for Plasma lipids, which measures total cholesterol, HDL cholesterol, LDL cholesterol, and triglycerides. Additionally these measures are used to calculate TC/HDL ratio.
Comprehensive Metabolic Panel | Four weeks
  A single venous blood sample will be collected and 200 ul added to a Piccolo test cartridge that measures glucose, creatinine, creatine kinase, blood urea nitrogen (BUN), total carbon dioxide, and chloride, sodium and potassium ions.

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany L Weir, PhD, Principal Investigator — Colorado State University
Locations (1):
- Colorado State University, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No